CLINICAL TRIAL: NCT06263933
Title: Effect of Experience Sharing and Mutual Assistance on Insight and Recovery During the First Psychotic Episode
Acronym: DIPEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Dominique JANUEL, head of research center and clinical professor, Centre hospitalier de Ville-Evrard, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01804-41
Record Dates: First submitted 2024-01-03; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-12

CONDITIONS: Psychotic Episode
Keywords: retablishment; insight; mutual assistance; peer helper; psychiatric hospitalization; first psychotic episode

STUDY DESIGN:
Intervention Model Description: A control group and a intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Patients are followed in routine care.
  Interventions: Other: Insight Scale; Other: Semi-directional interviews; Other: routine care
- DIPEM group (Experimental): Patients have 5 session of mutual assistance with a mediator psychologist, during five days, with 1 session per day. Each session lasts 1h30, with 45 min for atelier, 15 min for pause and 30 min about collective discussion.
  Interventions: Other: Insight Scale; Other: Semi-directional interviews; Other: session of mutual assistance with a mediator psychologist

INTERVENTIONS:
Other: Insight Scale — Before the patient was in DIPEM or control group and after the patient is involved in DIPEM or control group
  Other Names: stage of recovery scale
Other: Semi-directional interviews — In the end of the intervention. In the end of DIPEM Or in the end of control group.
  This intervention will be held after one month of hospitalization.
Other: routine care — routine care
  Arms: Control group
Other: session of mutual assistance with a mediator psychologist — session of mutual assistance with a mediator psychologist
  Arms: DIPEM group

SUMMARY:
Controlled, prospective, qualitative and quantitative trial. The goal of this trial is to evaluate the mutual assistance early intervention device efficacy and its impact on insight and personal recovery of participants living with a first psychotic episode. This intervention lasts 5 days with 1 session per day of 1 hour 30 minutes. Three evaluations, before the intervention, after intervention and 1 month after the hospitalization's end.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 40 years old
* First psychotic episode under the guidance of a doctor
* Brief psycotic trouble (SM-V)
* Presenting a first psychiatry hospitalization (all modalities hospitalizations combined)
* Fluent in French language (read and written)
* Patient affiliated to a social protection system or beneficiary of Medical Aid of State
* Patient having signed informed consent for his participation in the protocol

Exclusion Criteria:

* Patients whose clinical condition does not allow them to participate in research
* Patients placed in isolation rooms during the intervention

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-11-13 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
The level of the increasing of The INSIGHT scale | at baseline (T0) and at 5 days after the intervention's beginning (T1).
  Used the "Echelle de conscience de trouble" - insight scale. There are 8 items, with 3 choices for each items : agree, disagree, unsure. The time is 5 minutes.
  Maximum score = 12, very good Insight Minimum score= 0, No Insight 9 and more= good insight

SECONDARY OUTCOMES:
The increase of Recovery Scale | At baseline (T0) and at 5 days after the intervention's beginning (T1).
  Scale of recovery "Stage of recovery instrument" (STORI). The time is 25 minutes. There are 5 dimensions of recovery, with 10 groups of questions, with 50 items in total. There is 5 choices for each items, with "0" to "2" for "not at all true currently" and "3" to "5" is "completely true currently".
The semi-structured interview | At baseline (T0) and at 1 month after the hospitalization's end (T2).
  For the first semi-structured interview, with 11 questions on 3 themes : the crisis course and the hospitalization, the role of peers during hospitalization and finally afterwards hospitalization. For the second semi-structured interview, there are 13 questions with 4 themes : the hospitalization living, psychosocial functioning, trouble awareness and management of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Etablissement Public de Santé de Ville-Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andresen R, Oades L, Caputi P. The experience of recovery from schizophrenia: towards an empirically validated stage model. Aust N Z J Psychiatry. 2003 Oct;37(5):586-94. doi: 10.1046/j.1440-1614.2003.01234.x. PMID 14511087
- [Background] Courtet P. [Suicidal risk during the first psychotic episode]. Encephale. 2018 Dec;44(6S):S39-S43. doi: 10.1016/S0013-7006(19)30078-8. French. PMID 30935486
- [Background] Fennig S, Kovasznay B, Rich C, Ram R, Pato C, Miller A, Rubinstein J, Carlson G, Schwartz JE, Phelan J, et al. Six-month stability of psychiatric diagnoses in first-admission patients with psychosis. Am J Psychiatry. 1994 Aug;151(8):1200-8. doi: 10.1176/ajp.151.8.1200. PMID 8037256
- [Background] Franck N. [How to involve patients with schizophrenia in their treatment using psychoeducation]. Presse Med. 2016 Sep;45(9):742-8. doi: 10.1016/j.lpm.2016.07.012. Epub 2016 Aug 12. French. PMID 27526987
- [Background] Kessler RC, Amminger GP, Aguilar-Gaxiola S, Alonso J, Lee S, Ustun TB. Age of onset of mental disorders: a review of recent literature. Curr Opin Psychiatry. 2007 Jul;20(4):359-64. doi: 10.1097/YCO.0b013e32816ebc8c. PMID 17551351
- [Background] Malla A, McGorry P. Early Intervention in Psychosis in Young People: A Population and Public Health Perspective. Am J Public Health. 2019 Jun;109(S3):S181-S184. doi: 10.2105/AJPH.2019.305018. PMID 31242015
- [Background] Souaiby L, Gaillard R, Krebs MO. [Duration of untreated psychosis: A state-of-the-art review and critical analysis]. Encephale. 2016 Aug;42(4):361-6. doi: 10.1016/j.encep.2015.09.007. Epub 2016 May 6. French. PMID 27161262
- [Background] Thompson KN, McGorry PD, Harrigan SM. Reduced awareness of illness in first-episode psychosis. Compr Psychiatry. 2001 Nov-Dec;42(6):498-503. doi: 10.1053/comp.2001.27900. PMID 11704943